CLINICAL TRIAL: NCT00289588
Title: An Attempt to Reduce Community-Acquired Methicillin-Resistant Staphylococcus Aureus Infection in Soldiers: a Controlled Trial
Brief Title: An Attempt to Reduce Community-Acquired Methicillin-Resistant Staphylococcus Aureus (MRSA) Infection in Soldiers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Becton, Dickinson and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C.2004.163
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2005-12

CONDITIONS: Community-Acquired MRSA Infections; Abscesses; Cellulitis; Folliculitis
Keywords: Methicillin-resistant Staphylococcus aureus; Staphylococcus aureus; MRSA; CA-MRSA
MeSH Terms: conditions — Abscess; Cellulitis; Folliculitis; Staphylococcal Infections | interventions — Mupirocin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Mupirocin (drug)

SUMMARY:
The main purpose of this study is to determine if applying mupirocin into soldiers noses who are colonized with methicillin-resistant Staphylococcus aureus (MRSA) will reduce infections in them and their cohort of fellow soldiers.

DETAILED DESCRIPTION:
Community-acquired MRSA infections are increasingly common in the community and in particular among certain groups of which soldiers are one. Many researchers and clinicians have postulated that one method to prevent infections is to selectively eradicate CA-MRSA in those who are colonized with the pathogen. The two main purposes of the study are: to determine if selective CA-MRSA eradication in subjects reduces infections in the CA-MRSA colonized individual; and to determine if selective CA-MRSA eradication in subjects reduces infections in the study cohort. Other information concerning CA-MRSA includes: prevalence, risk factors, and virulence data. The population will be soldiers enrolled in the combat medic training class at Ft. Sam Houston. We will enroll approximately 3000 soldiers over a two year period. After informed written consent, we will culture their anterior nares nares and administer questionnaires at the beginning and at the end of the study, following them prospectively for infections. The follow-up period will be 16 weeks. For those with CA-MRSA in their nares, they will be randomized (by cohort) to receive either 5 days of mupirocin or placebo.

ELIGIBILITY:
Inclusion Criteria:Soldiers enrolled into the combat medic course at Ft. Sam Houston, TX.

-

Exclusion Criteria: Allergy to mupirocin.

-

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000
Dates: Start 2005-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Soft tissue infections in subjects who received the study medication and soft tissue infections in the study cohorts.

SECONDARY OUTCOMES:
Changes in S. aureus carriage rates (including MRSA).

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Ellis, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Ellis MW, Hospenthal DR, Dooley DP, Gray PJ, Murray CK. Natural history of community-acquired methicillin-resistant Staphylococcus aureus colonization and infection in soldiers. Clin Infect Dis. 2004 Oct 1;39(7):971-9. doi: 10.1086/423965. Epub 2004 Sep 2. PMID 15472848